CLINICAL TRIAL: NCT00327873
Title: A Multi-center Randomized Double-blind Controlled Trial of Oxygen Versus Medical Air for the Relief of Breathlessness in Patients With Intractable Dyspnea and PaO2>55mmHg
Brief Title: Palliative Oxygen for the Relief of Breathlessness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Health and Medical Research Council, Australia (Other)
Collaborators: Doris Duke Charitable Foundation (Other); Cancer Council Tasmania (Other); Duke Institute on Care at the End of Life, USA (Unknown); Flinders Medical Research Institute Small Research Grants Scheme, Australia (Unknown)
Responsible Party: Amy Abernethy, MD, Assistant Professor of Medicine, Duke Cancer Care Research Program, Duke University Medical Center
Organization: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AG0064
Record Dates: First submitted 2006-05-18; First posted 2006-05-19 (Estimated); Last update posted 2009-12-14 (Estimated); Status verified 2009-02

CONDITIONS: Dyspnea
Keywords: breathlessness; shortness of breath; end-of-life care; hospice
MeSH Terms: conditions — Dyspnea | interventions — Oxygen; Air

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Oxygen
  Interventions: Other: Oxygen
- B (Active Comparator): Medical Air
  Interventions: Other: Medical Air

INTERVENTIONS:
Other: Oxygen — 2L/min for 15 hours or greater per day via concentrator and nasal cannulae for 7 days
  Arms: A
Other: Medical Air — 2L/min for 15 hours or greater per day via concentrator and nasal cannulae for 7 days
  Arms: B

SUMMARY:
The main goal of this study is to establish the effectiveness of palliative oxygen in the context within which it is usually provided--relief of the sensation of breathlessness and improvement in quality of life for people with maximally-treated life-limiting illness.

DETAILED DESCRIPTION:
When further medical management will not relieve intractable breathlessness, palliative oxygen is often prescribed regardless of whether the person meets the common oxygen funding criteria of severely low blood oxygen levels. The results of this study will inform best practice in the care of people with advanced life-limiting illness and intractable breathlessness, aid in the development of rational funding guidelines, and answer an international debate on the role of palliative oxygen.

This study is a definitive international multi-center randomized double-blind controlled trial of oxygen versus medical air for the relief of breathlessness in participants with intractable dyspnea and PaO2>55mmHg (a measure of blood oxygen levels). Specific aims include demonstration of the effectiveness of oxygen versus medical air in relieving breathlessness in the palliative setting (Specific Aim 1) and improving QOL (Specific Aim 2). Additionally, we will seek to establish which patients derive the greatest benefit (Specific Aim 3), the risks of therapy (Specific Aim 4), and the costs of therapy (Specific Aim 5). The primary hypothesis is that oxygen therapy is superior to air in relieving the sensation of breathlessness for patients with intractable dyspnea due to life-limiting illness in the setting of PaO2>55mmHg.

All participants are enrolled as outpatients. The "eligibility visit" occurs about 5-7 days before starting the study and will include review of the consent form, a short interview, physical exam, and blood tests. The visit can occur in the home or clinic. The blood tests include regular venipuncture and also an arterial blood gas, if these studies have not been done in the preceding month. The "randomization visit" occurs 2 days before the study starts (Day -2) and includes a short interview and quality of life (QOL) questionnaire; this visit is usually done in the home but can also occur in the clinic. The oxygen or air concentrators are delivered to the home on Day 0 by a trained person from the oxygen company. On the same day there is also a brief home visit from the study nurse that includes a short interview and QOL questionnaire. The participant uses the oxygen or medical air gas each of 7 days (Days 0-6) for at least 15 hours each day. While using the oxygen/air the participant fills out a short diary form in the morning and evening, within 30 minutes of waking up or retiring. The diary focuses on the breathlessness, how the participant is feeling, and potential side effects of the gas. The study nurse conducts a "check-in" telephone call on Day 3 to make sure the participant is doing OK. On the last day (Day 6) the nurse visits the home to conduct a brief interview with a short QOL questionnaire. The oxygen company will pick up the concentrator, usually on Day 7.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with intractable dyspnea and PaO2>55mmHg in the setting of terminal illness where the underlying cause has been maximally treated; a medical specialist must document that all identified reversible causes of the dyspnea have been treated; PaO2 measurement must be in the last month
* Dyspnea at rest or with minimal exertion, as measured by a score of ≥ 3 on the Medical Research Council categorical dyspnea exertion scale
* On stable medications over the prior week except routine "as needed" medications.
* Survival of at least 1 month in the opinion of the treating physician

Exclusion Criteria:

* Meets international guidelines for long-term oxygen therapy with PaO2 56-59mmHg, i.e. symptomatic pulmonary hypertension with cor pulmonale
* Hemoglobin<10.0g/dL as measured within one month of baseline evaluation
* PaCO2 >50 mm Hg.
* Confusion as measured by Folstein Mini-mental Status Exam <24/30
* Current oxygen therapy or continuous oxygen therapy in previous week
* Actively smoking
* Active respiratory or cardiac event in the previous 2 weeks, not including upper respiratory tract infections; illness must be resolved for at least 2 weeks prior to baseline evaluation, as judged by a doctor involved in the care of the patient
* Previous respiratory failure induced by oxygen
* Unable to give informed consent or complete diary entries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2005-05; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Changes in relief from the sensation of breathlessness | 7 days

SECONDARY OUTCOMES:
Changes in quality of life (QOL) | 7 days
Identification of patients who benefit from palliative oxygen | 7 days
Identification of side effects | 7 days
Documentation of costs of palliative oxygen | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Amy Abernethy, MD, Principal Investigator — Duke University; David Curow, BMed,FRACP,MPH, Principal Investigator — Flinders University, Australia
Locations (7):
- Duke University Department of Medicine, Division of Medical Oncology, Durham, North Carolina, United States
- Australia (4):
  - Sydney Area Health Service, Sydney Cancer Centre, Sydney, New South Wales
  - Flinders University, Southern Adelaide Palliative Services, Adelaide, South Australia
  - Statewide Palliative Care Service, Launceston, Tasmania
  - Austin Health, Melbourne, Victoria
- United Kingdom (2):
  - St Nicholas Hospice, Cambridge, Cambridge
  - Nottingham University, Nottingham, Nottingham

REFERENCES:
- [Background] Abernethy AP, Currow DC, Frith P, Fazekas B. Prescribing palliative oxygen: a clinician survey of expected benefit and patterns of use. Palliat Med. 2005 Mar;19(2):168-70. doi: 10.1177/026921630501900219. No abstract available. PMID 15810762
- [Background] Booth S, Wade R, Johnson M, Kite S, Swannick M, Anderson H; Expert Working Group of the Scientific Committee of the Association of Palliative Medicine. The use of oxygen in the palliation of breathlessness. A report of the expert working group of the Scientific Committee of the Association of Palliative Medicine. Respir Med. 2004 Jan;98(1):66-77. doi: 10.1016/j.rmed.2003.08.008. PMID 14959816
- [Background] Guyatt GH, McKim DA, Austin P, Bryan R, Norgren J, Weaver B, Goldstein RS. Appropriateness of domiciliary oxygen delivery. Chest. 2000 Nov;118(5):1303-8. doi: 10.1378/chest.118.5.1303. PMID 11083678
- [Background] Bruera E, Sweeney C, Willey J, Palmer JL, Strasser F, Morice RC, Pisters K. A randomized controlled trial of supplemental oxygen versus air in cancer patients with dyspnea. Palliat Med. 2003 Dec;17(8):659-63. doi: 10.1191/0269216303pm826oa. PMID 14694916
- [Derived] Abernethy AP, McDonald CF, Frith PA, Clark K, Herndon JE 2nd, Marcello J, Young IH, Bull J, Wilcock A, Booth S, Wheeler JL, Tulsky JA, Crockett AJ, Currow DC. Effect of palliative oxygen versus room air in relief of breathlessness in patients with refractory dyspnoea: a double-blind, randomised controlled trial. Lancet. 2010 Sep 4;376(9743):784-93. doi: 10.1016/S0140-6736(10)61115-4. PMID 20816546
- See also: ISRCTN67448752 on Current Controlled Trials — http://www.controlled-trials.com/ISRCTN67448752/ISRCTN67448752